CLINICAL TRIAL: NCT00003511
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Multiple Myeloma
Brief Title: Antineoplaston Therapy in Treating Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066554; BC-MM-2 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: Stage I multiple myeloma; Stage II multiple myeloma; Stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Multiple Myeloma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Multiple Myeloma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Multiple Myeloma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Multiple Myeloma.

DETAILED DESCRIPTION:
Multiple Myeloma patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Multiple Myeloma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Multiple Myeloma.
* To determine objective response, tumor size is measured utilizing physical examination, radiologic studies, and bone marrow biopsies as necessary, performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and biochemically confirmed recurrent or progressing multiple myeloma that is unlikely to respond to existing therapy, including surgery, radiotherapy, and chemotherapy

  * At least one standard first line therapy failure
* No localized plasmacytoma or plasmacytosis limited to the bone marrow
* Evidence of tumor by MRI or CT scan
* Presence of myeloma proteins in serum and urine, including Bence-Jones proteins

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic insufficiency

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal problems
* No renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No serious medical or psychiatric disorders
* No active infections

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered (patients with multiple tumors who have received radiotherapy to some, but not all, tumors may be admitted earlier than 8 weeks)

Surgery:

* Must be recovered from prior surgery

Other:

* Prior cytodifferentiating agent allowed
* No prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1996-04-04 (Actual); Primary Completion 1999-10-21 (Actual); Study Completion 1999-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with Multiple Myeloma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 5
Completed | 1
Not Completed | 4
Not completed — Not evaluable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 51.2 [43.8 to 75.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response, Stable Disease, Progressive Disease or Not Evaluable
Description: Objective response rate per The International Working Group response criteria (1999): Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least four weeks. Stable Disease (SD), < 50% change in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least twelve weeks.
Time Frame: 36 months
Population: All patients enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 5
participants
  Objective response | 0
  Stable Disease | 1
  Progressive Disease | 0
  Not evaluable | 4

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=5)
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Pain: Pelvis (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=5)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 3
Hypertension (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Non-functional Central Venous Catheter (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Fever (General disorders) | 1
Weight gain (General disorders) | 1
Edema/Fluid retention (Skin and subcutaneous tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2
Nausea (General disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage, GU (Renal and urinary disorders) | 1
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 2
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Alkaline phosphatase (Infections and infestations) | 1
Hyperglycemia (Investigations) | 1
Hypernatremia (Investigations) | 3
Hypocalcemia (Investigations) | 2
Hypokalemia (Investigations) | 2
Hypomagnesemia (Investigations) | 1
SGOT (Investigations) | 1
Uric acid, serum-high (hyperuricemia) (Investigations) | 2
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 2
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Pelvis (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (shortness of breath) (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No